CLINICAL TRIAL: NCT05973994
Title: Shockwave Induced Attenuation of Calcified Plaques Quantified With OCT
Acronym: SCALPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Prof. Giuseppe Sangiorgi, Professor, University of Rome Tor Vergata
Other Study IDs: 75/21
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Calcification
Keywords: Coronary artery calcification; Intravascular Lithotripsy; Optical Coherence Tomography; Calcium density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with significant calcific coronary artery stenosis candidate to PCI: Patients with coronary artery calcifications responsible for significant stenosis will undergo basal OCT acquistion. After intravascular lithotripsy (IVL) application, a second OCT acquisition will be made. The mean calcium density of the vessel's ROI before IVL and after IVL will be compared. Stent implantation will be performed after the second OCT acquisition.
  Interventions: Device: intravascular lithotripsy with Shockwave coronary system

INTERVENTIONS:
Device: intravascular lithotripsy with Shockwave coronary system — OCT acquistion is performed at baseline. Then the IVL catheter will be passed across the lesion over the guidewire. Atherectomy or cutting/scoring balloons is not permitted per protocol. The IVL procedure is considered successful when a residual stenosis <50% by visual estimate after IVL alone is achieved. After IVL procedure, one OCT imaging acquisition must be performed. If the residual stenosis is ≥50% following IVL, noncompliant balloon dilatation will be performed prior to stenting and OCT images repeated accordingly. Subsequent stent implantation will be performed per local standard of care at the discretion of the operator. Following stent implantation, high pressure post-dilatation is recommended and OCT imaging acquisition must be performed to assess stent apposition for secondary end point.
  Other Names: OCT acquisition with FD-OCT imaging catheter

SUMMARY:
The goal of this observational, prospective, multicenter study is to explore local action of coronary calcium fragmentation exerted by endovascular lithotripsy by images acquired with OCT, in patients with coronary artery calcifications responsible for significant stenosis, candidate to PCI. The main question it aims to answer, is the ability of Shockwave System to reduce calcium density in the Region of Interest (ROI) of the vessel wall.

DETAILED DESCRIPTION:
Coronary arteries with calcific lesions will undergo intravasculary lithotripsy (IVL) treatment; OCT acquisition will be performed before IVL treatment, after IVL treatment and after stent-implantation. All OCT frames will be uploaded on the image processing and analysis program ImageJ (US National Institutes of Health). ROI will be selected as part of image where calcium is located. Image analysis will be performed using frequency histogram of pixel density in the ROI pre- and post-IVL, as a measure of calcium density. Mean pixel density of the ROI before IVL will be compared with mean pixel density of the ROI after IVL, measuring delta pixel density.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI
* Left ventricular ejection fraction (LVEF) ≥35% as measured prior to enrollment
* eGFR ≥45 ml/min (Cockroft-Gault, MDRD)
* Troponin must be less than or equal to the upper limit of lab normal value within 24 hours prior to the procedure or if troponin is elevated, concomitant CK must be normal
* Ability to tolerate dual antiplatelet therapy (i.e. aspirin and clopidogrel, prasugrel, or ticagrelor) for at least 6 months (for patient not on oral anticoagulation) and single antiplatelet therapy for life
* The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
* Single de novo target lesion stenosis of LAD, RCA or LCX (or of their branches) with stenosis of ≥70% and <100% or stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80, or iFR <0.89 or IVUS or OCT minimum lumen area ≤4.0 mm²
* Reference vessel must have 2.5 mm - 4.0 mm diameter and ≤ 30 mm length
* Evidence of calcification at the lesion site assessed by angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, or by IVUS or OCT, with presence of ≥270 degrees of calcium on at least 1 cross section
* Planned treatment of single lesion for every target vessel
* Ability to pass a 0.014" guide wire across the lesion
* The target vessel must have a TIMI flow 3 at baseline

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) <35%
* Subject is pregnant or nursing
* eGFR <45 ml/min (Cockroft-Gault, MDRD) or chronic dialysis
* Untreated pre-procedural haemoglobin <9 g/dL or intention to refuse blood transfusions if one should become necessary
* Patient has a platelet count <100,000 cells/mm3 or >750,000 cells/mm3
* Patient has a known allergy to protocol required medications (clopidogrel, thienopyridines, aspirin, contrast media) that cannot be adequately premedicated
* Uncontrolled diabetes defined as a fasting hyperglycaemia >200 mg/dL or HbA1c greater than or equal to 10%
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Patient has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Patient has a history of coagulopathy
* Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint
* Subjects with a life expectancy of less than 1 year
* Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
* Planned use of atherectomy, scoring or cutting balloon, or any investigational device other than lithotripsy
* Stent implantation in the target vessel within the last year or a stent within 10 mm of the target lesion
* Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel
* Angiographic evidence of a dissection in the target vessel at baseline or after guidewire passage

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the Catheterization Laboratory that undergo coronary angiography, are potentially selected.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of calcium density in the Region of Interest (ROI) of the vessel after lithotripsy treatment | five-ten minutes
  Calcium density is measured as delta pixel-density between calcific lesions images before and after lithotripsy at OCT acquisition

SECONDARY OUTCOMES:
Reduction of stent malapposition after intracoronary lithotripsy application | five minutes after stent impantation
  Sten malapposition is measured as the distance between the abluminal surface of the strut and the luminal surface of the artery wall in the frames of lesion acquired by OCT after stent implantation.
Incidence of acute vessel dissection and acute stent thrombosis or subacute vessel thrombosis after index procedure | one, six months
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe M Sangiorgi, Professor, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- University of Rome Tor Vergata - Policlinico, Roma, Rome, Italy

REFERENCES:
- [Background] Abdel-Wahab M, Richardt G, Joachim Buttner H, Toelg R, Geist V, Meinertz T, Schofer J, King L, Neumann FJ, Khattab AA. High-speed rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: the randomized ROTAXUS (Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2013 Jan;6(1):10-9. doi: 10.1016/j.jcin.2012.07.017. Epub 2012 Dec 19. PMID 23266232
- [Background] Agarwal S, Cox AJ, Herrington DM, Jorgensen NW, Xu J, Freedman BI, Carr JJ, Bowden DW. Coronary calcium score predicts cardiovascular mortality in diabetes: diabetes heart study. Diabetes Care. 2013 Apr;36(4):972-7. doi: 10.2337/dc12-1548. Epub 2012 Dec 10. PMID 23230101
- [Background] Ali ZA, Brinton TJ, Hill JM, Maehara A, Matsumura M, Karimi Galougahi K, Illindala U, Gotberg M, Whitbourn R, Van Mieghem N, Meredith IT, Di Mario C, Fajadet J. Optical Coherence Tomography Characterization of Coronary Lithoplasty for Treatment of Calcified Lesions: First Description. JACC Cardiovasc Imaging. 2017 Aug;10(8):897-906. doi: 10.1016/j.jcmg.2017.05.012. PMID 28797412
- [Background] Ali ZA, Nef H, Escaned J, Werner N, Banning AP, Hill JM, De Bruyne B, Montorfano M, Lefevre T, Stone GW, Crowley A, Matsumura M, Maehara A, Lansky AJ, Fajadet J, Di Mario C. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10):e008434. doi: 10.1161/CIRCINTERVENTIONS.119.008434. Epub 2019 Sep 25. PMID 31553205
- [Background] Allison MA, Criqui MH, Wright CM. Patterns and risk factors for systemic calcified atherosclerosis. Arterioscler Thromb Vasc Biol. 2004 Feb;24(2):331-6. doi: 10.1161/01.ATV.0000110786.02097.0c. Epub 2003 Dec 4. PMID 14656730
- [Background] Barbato E, Shlofmitz E, Milkas A, Shlofmitz R, Azzalini L, Colombo A. State of the art: evolving concepts in the treatment of heavily calcified and undilatable coronary stenoses - from debulking to plaque modification, a 40-year-long journey. EuroIntervention. 2017 Aug 25;13(6):696-705. doi: 10.4244/EIJ-D-17-00473. PMID 28844031
- [Background] Baumbach A, Bittl JA, Fleck E, Geschwind HJ, Sanborn TA, Tcheng JE, Karsch KR. Acute complications of excimer laser coronary angioplasty: a detailed analysis of multicenter results. Coinvestigators of the U.S. and European Percutaneous Excimer Laser Coronary Angioplasty (PELCA) Registries. J Am Coll Cardiol. 1994 May;23(6):1305-13. doi: 10.1016/0735-1097(94)90371-9. PMID 8176087
- [Background] Benezet J, Diaz de la Llera LS, Cubero JM, Villa M, Fernandez-Quero M, Sanchez-Gonzalez A. Drug-eluting stents following rotational atherectomy for heavily calcified coronary lesions: long-term clinical outcomes. J Invasive Cardiol. 2011 Jan;23(1):28-32. PMID 21183767
- [Background] Bhatt P, Parikh P, Patel A, Chag M, Chandarana A, Parikh R, Parikh K. Long-term safety and performance of the orbital atherectomy system for treating calcified coronary artery lesions: 5-Year follow-up in the ORBIT I trial. Cardiovasc Revasc Med. 2015 Jun;16(4):213-6. doi: 10.1016/j.carrev.2015.03.007. Epub 2015 Mar 31. PMID 25866032
- [Background] Bourantas CV, Zhang YJ, Garg S, Iqbal J, Valgimigli M, Windecker S, Mohr FW, Silber S, Vries Td, Onuma Y, Garcia-Garcia HM, Morel MA, Serruys PW. Prognostic implications of coronary calcification in patients with obstructive coronary artery disease treated by percutaneous coronary intervention: a patient-level pooled analysis of 7 contemporary stent trials. Heart. 2014 Aug;100(15):1158-64. doi: 10.1136/heartjnl-2013-305180. Epub 2014 May 20. PMID 24846971
- [Background] Brinton TJ, Ali ZA, Hill JM, Meredith IT, Maehara A, Illindala U, Lansky A, Gotberg M, Van Mieghem NM, Whitbourn R, Fajadet J, Di Mario C. Feasibility of Shockwave Coronary Intravascular Lithotripsy for the Treatment of Calcified Coronary Stenoses. Circulation. 2019 Feb 5;139(6):834-836. doi: 10.1161/CIRCULATIONAHA.118.036531. No abstract available. PMID 30715944
- [Background] Brodmann M, Holden A, Zeller T. Safety and Feasibility of Intravascular Lithotripsy for Treatment of Below-the-Knee Arterial Stenoses. J Endovasc Ther. 2018 Aug;25(4):499-503. doi: 10.1177/1526602818783989. Epub 2018 Jun 18. PMID 29911480
- [Background] Brodmann M, Werner M, Brinton TJ, Illindala U, Lansky A, Jaff MR, Holden A. Safety and Performance of Lithoplasty for Treatment of Calcified Peripheral Artery Lesions. J Am Coll Cardiol. 2017 Aug 15;70(7):908-910. doi: 10.1016/j.jacc.2017.06.022. No abstract available. PMID 28797363
- [Background] Brodmann M, Werner M, Holden A, Tepe G, Scheinert D, Schwindt A, Wolf F, Jaff M, Lansky A, Zeller T. Primary outcomes and mechanism of action of intravascular lithotripsy in calcified, femoropopliteal lesions: Results of Disrupt PAD II. Catheter Cardiovasc Interv. 2019 Feb 1;93(2):335-342. doi: 10.1002/ccd.27943. Epub 2018 Nov 25. PMID 30474206
- [Background] Budoff MJ, Young R, Burke G, Jeffrey Carr J, Detrano RC, Folsom AR, Kronmal R, Lima JAC, Liu KJ, McClelland RL, Michos E, Post WS, Shea S, Watson KE, Wong ND. Ten-year association of coronary artery calcium with atherosclerotic cardiovascular disease (ASCVD) events: the multi-ethnic study of atherosclerosis (MESA). Eur Heart J. 2018 Jul 1;39(25):2401-2408. doi: 10.1093/eurheartj/ehy217. PMID 29688297
- [Background] Busse A, Cantre D, Beller E, Streckenbach F, Oner A, Ince H, Weber MA, Meinel FG. Cardiac CT: why, when, and how : Update 2019. Radiologe. 2019 Dec;59(Suppl 1):1-9. doi: 10.1007/s00117-019-0530-9. PMID 31062037
- [Background] Chambers JW, Feldman RL, Himmelstein SI, Bhatheja R, Villa AE, Strickman NE, Shlofmitz RA, Dulas DD, Arab D, Khanna PK, Lee AC, Ghali MG, Shah RR, Davis TP, Kim CY, Tai Z, Patel KC, Puma JA, Makam P, Bertolet BD, Nseir GY. Pivotal trial to evaluate the safety and efficacy of the orbital atherectomy system in treating de novo, severely calcified coronary lesions (ORBIT II). JACC Cardiovasc Interv. 2014 May;7(5):510-8. doi: 10.1016/j.jcin.2014.01.158. PMID 24852804
- [Background] Chen NX, Moe SM. Vascular calcification: pathophysiology and risk factors. Curr Hypertens Rep. 2012 Jun;14(3):228-37. doi: 10.1007/s11906-012-0265-8. PMID 22476974
- [Background] Choi KH, Song YB, Lee JM, Lee SY, Park TK, Yang JH, Choi JH, Choi SH, Gwon HC, Hahn JY. Impact of Intravascular Ultrasound-Guided Percutaneous Coronary Intervention on Long-Term Clinical Outcomes in Patients Undergoing Complex Procedures. JACC Cardiovasc Interv. 2019 Apr 8;12(7):607-620. doi: 10.1016/j.jcin.2019.01.227. Epub 2019 Mar 13. PMID 30878474
- [Background] Costopoulos C, Naganuma T, Colombo A. Tools and techniques clinical: percutaneous intervention of calcific coronary lesions. EuroIntervention. 2014 Jan 22;9(9):1124-6. doi: 10.4244/EIJV9I9A188. No abstract available. PMID 24457284
- [Background] de Ribamar Costa J Jr, Mintz GS, Carlier SG, Mehran R, Teirstein P, Sano K, Liu X, Lui J, Na Y, Castellanos C, Biro S, Dani L, Rinker J, Moussa I, Dangas G, Lansky AJ, Kreps EM, Collins M, Stone GW, Moses JW, Leon MB. Nonrandomized comparison of coronary stenting under intravascular ultrasound guidance of direct stenting without predilation versus conventional predilation with a semi-compliant balloon versus predilation with a new scoring balloon. Am J Cardiol. 2007 Sep 1;100(5):812-7. doi: 10.1016/j.amjcard.2007.03.100. Epub 2007 Jun 13. PMID 17719325
- [Background] de Waha S, Allali A, Buttner HJ, Toelg R, Geist V, Neumann FJ, Khattab AA, Richardt G, Abdel-Wahab M. Rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: Two-year clinical outcome of the randomized ROTAXUS trial. Catheter Cardiovasc Interv. 2016 Mar;87(4):691-700. doi: 10.1002/ccd.26290. Epub 2015 Nov 3. PMID 26525804
- [Background] Demer LL, Tintut Y. Vascular calcification: pathobiology of a multifaceted disease. Circulation. 2008 Jun 3;117(22):2938-48. doi: 10.1161/CIRCULATIONAHA.107.743161. No abstract available. PMID 18519861
- [Background] di Mario C, Koskinas KC, Raber L. Clinical Benefit of IVUS Guidance for Coronary Stenting: The ULTIMATE Step Toward Definitive Evidence? J Am Coll Cardiol. 2018 Dec 18;72(24):3138-3141. doi: 10.1016/j.jacc.2018.10.029. No abstract available. PMID 30545452
- [Background] Di Mario C, Ramasami N. Techniques to enhance guide catheter support. Catheter Cardiovasc Interv. 2008 Oct 1;72(4):505-12. doi: 10.1002/ccd.21670. No abstract available. PMID 18814225
- [Background] Dini CS, Tomberli B, Mattesini A, Ristalli F, Valente S, Stolcova M, Meucci F, Baldereschi G, Fanelli F, Shlofmitz RA, Ali ZA, Di Mario C. Intravascular lithotripsy for calcific coronary and peripheral artery stenoses. EuroIntervention. 2019 Oct 20;15(8):714-721. doi: 10.4244/EIJ-D-18-01056. PMID 31062700
- [Background] Dippel EJ, Kereiakes DJ, Tramuta DA, Broderick TM, Shimshak TM, Roth EM, Hattemer CR, Runyon JP, Whang DD, Schneider JF, Abbottsmith CW. Coronary perforation during percutaneous coronary intervention in the era of abciximab platelet glycoprotein IIb/IIIa blockade: an algorithm for percutaneous management. Catheter Cardiovasc Interv. 2001 Mar;52(3):279-86. doi: 10.1002/ccd.1065. PMID 11246236
- [Background] Faggiano P, Dasseni N, Gaibazzi N, Rossi A, Henein M, Pressman G. Cardiac calcification as a marker of subclinical atherosclerosis and predictor of cardiovascular events: A review of the evidence. Eur J Prev Cardiol. 2019 Jul;26(11):1191-1204. doi: 10.1177/2047487319830485. Epub 2019 Mar 7. PMID 30845832
- [Background] Fourrier JL, Bertrand ME, Auth DC, Lablanche JM, Gommeaux A, Brunetaud JM. Percutaneous coronary rotational angioplasty in humans: preliminary report. J Am Coll Cardiol. 1989 Nov 1;14(5):1278-82. doi: 10.1016/0735-1097(89)90428-2. PMID 2808983
- [Background] Friedrich GJ, Moes NY, Muhlberger VA, Gabl C, Mikuz G, Hausmann D, Fitzgerald PJ, Yock PG. Detection of intralesional calcium by intracoronary ultrasound depends on the histologic pattern. Am Heart J. 1994 Sep;128(3):435-41. doi: 10.1016/0002-8703(94)90614-9. PMID 8074002
- [Background] Fujino A, Mintz GS, Matsumura M, Lee T, Kim SY, Hoshino M, Usui E, Yonetsu T, Haag ES, Shlofmitz RA, Kakuta T, Maehara A. A new optical coherence tomography-based calcium scoring system to predict stent underexpansion. EuroIntervention. 2018 Apr 6;13(18):e2182-e2189. doi: 10.4244/EIJ-D-17-00962. PMID 29400655
- [Background] Genereux P, Lee AC, Kim CY, Lee M, Shlofmitz R, Moses JW, Stone GW, Chambers JW. Orbital Atherectomy for Treating De Novo Severely Calcified Coronary Narrowing (1-Year Results from the Pivotal ORBIT II Trial). Am J Cardiol. 2015 Jun 15;115(12):1685-90. doi: 10.1016/j.amjcard.2015.03.009. Epub 2015 Mar 24. PMID 25910525
- [Background] Greenland P, LaBree L, Azen SP, Doherty TM, Detrano RC. Coronary artery calcium score combined with Framingham score for risk prediction in asymptomatic individuals. JAMA. 2004 Jan 14;291(2):210-5. doi: 10.1001/jama.291.2.210. PMID 14722147
- [Background] Guedeney P, Claessen BE, Mehran R, Mintz GS, Liu M, Sorrentino S, Giustino G, Farhan S, Leon MB, Serruys PW, Smits PC, von Birgelen C, Ali ZA, Genereux P, Redfors B, Madhavan MV, Ben-Yehuda O, Stone GW. Coronary Calcification and Long-Term Outcomes According to Drug-Eluting Stent Generation. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1417-1428. doi: 10.1016/j.jcin.2020.03.053. PMID 32553329
- [Background] Hill JM, Kereiakes DJ, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646. doi: 10.1016/j.jacc.2020.09.603. Epub 2020 Oct 15. PMID 33069849
- [Background] Hoffmann R, Mintz GS, Popma JJ, Satler LF, Kent KM, Pichard AD, Leon MB. Treatment of calcified coronary lesions with Palmaz-Schatz stents. An intravascular ultrasound study. Eur Heart J. 1998 Aug;19(8):1224-31. doi: 10.1053/euhj.1998.1028. PMID 9740344
- [Background] Hofmann Bowman MA, McNally EM. Genetic pathways of vascular calcification. Trends Cardiovasc Med. 2012 May;22(4):93-8. doi: 10.1016/j.tcm.2012.07.002. PMID 23040839
- [Background] Hong SJ, Mintz GS, Ahn CM, Kim JS, Kim BK, Ko YG, Kang TS, Kang WC, Kim YH, Hur SH, Hong BK, Choi D, Kwon H, Jang Y, Hong MK; IVUS-XPL Investigators. Effect of Intravascular Ultrasound-Guided Drug-Eluting Stent Implantation: 5-Year Follow-Up of the IVUS-XPL Randomized Trial. JACC Cardiovasc Interv. 2020 Jan 13;13(1):62-71. doi: 10.1016/j.jcin.2019.09.033. PMID 31918944
- [Background] Huisman J, van der Heijden LC, Kok MM, Louwerenburg JH, Danse PW, Jessurun GA, de Man FH, Lowik MM, Linssen GC, IJzerman MJ, Doggen CJ, von Birgelen C. Two-year outcome after treatment of severely calcified lesions with newer-generation drug-eluting stents in acute coronary syndromes: A patient-level pooled analysis from TWENTE and DUTCH PEERS. J Cardiol. 2017 Apr;69(4):660-665. doi: 10.1016/j.jjcc.2016.06.010. Epub 2016 Jul 28. PMID 27476343
- [Background] Johnson RC, Leopold JA, Loscalzo J. Vascular calcification: pathobiological mechanisms and clinical implications. Circ Res. 2006 Nov 10;99(10):1044-59. doi: 10.1161/01.RES.0000249379.55535.21. PMID 17095733
- [Background] Kalra SS, Shanahan CM. Vascular calcification and hypertension: cause and effect. Ann Med. 2012 Jun;44 Suppl 1:S85-92. doi: 10.3109/07853890.2012.660498. PMID 22713153
- [Background] Kassimis G, Raina T, Kontogiannis N, Patri G, Abramik J, Zaphiriou A, Banning AP. How Should We Treat Heavily Calcified Coronary Artery Disease in Contemporary Practice? From Atherectomy to Intravascular Lithotripsy. Cardiovasc Revasc Med. 2019 Dec;20(12):1172-1183. doi: 10.1016/j.carrev.2019.01.010. Epub 2019 Jan 10. PMID 30711477
- [Background] Kawamoto H, Latib A, Ruparelia N, Boccuzzi GG, Pennacchi M, Sardella G, Garbo R, Meliga E, D'Ascenzo F, Moretti C, Rossi ML, Presbitero P, Ielasi A, Magri C, Nakamura S, Colombo A. Planned versus provisional rotational atherectomy for severe calcified coronary lesions: Insights From the ROTATE multi-center registry. Catheter Cardiovasc Interv. 2016 Nov 15;88(6):881-889. doi: 10.1002/ccd.26411. Epub 2016 Jan 17. PMID 26775275
- [Background] Kawasaki M, Bouma BE, Bressner J, Houser SL, Nadkarni SK, MacNeill BD, Jang IK, Fujiwara H, Tearney GJ. Diagnostic accuracy of optical coherence tomography and integrated backscatter intravascular ultrasound images for tissue characterization of human coronary plaques. J Am Coll Cardiol. 2006 Jul 4;48(1):81-8. doi: 10.1016/j.jacc.2006.02.062. Epub 2006 Jun 9. PMID 16814652
- [Background] Kereiakes DJ, Hill JM, Ben-Yehuda O, Maehara A, Alexander B, Stone GW. Evaluation of safety and efficacy of coronary intravascular lithotripsy for treatment of severely calcified coronary stenoses: Design and rationale for the Disrupt CAD III trial. Am Heart J. 2020 Jul;225:10-18. doi: 10.1016/j.ahj.2020.04.005. Epub 2020 Apr 18. PMID 32470635
- [Background] Kini AS, Vengrenyuk Y, Pena J, Motoyama S, Feig JE, Meelu OA, Rajamanickam A, Bhat AM, Panwar S, Baber U, Sharma SK. Optical coherence tomography assessment of the mechanistic effects of rotational and orbital atherectomy in severely calcified coronary lesions. Catheter Cardiovasc Interv. 2015 Nov 15;86(6):1024-32. doi: 10.1002/ccd.26000. Epub 2015 May 11. PMID 25964009
- [Background] Kobayashi Y, Okura H, Kume T, Yamada R, Kobayashi Y, Fukuhara K, Koyama T, Nezuo S, Neishi Y, Hayashida A, Kawamoto T, Yoshida K. Impact of target lesion coronary calcification on stent expansion. Circ J. 2014;78(9):2209-14. doi: 10.1253/circj.cj-14-0108. Epub 2014 Jul 14. PMID 25017740
- [Background] Kurbaan AS, Kelly PA, Sigwart U. Cutting balloon angioplasty and stenting for aorto-ostial lesions. Heart. 1997 Apr;77(4):350-2. doi: 10.1136/hrt.77.4.350. PMID 9155615
- [Background] Lee MS, Shlofmitz E, Kaplan B, Alexandru D, Meraj P, Shlofmitz R. Real-World Multicenter Registry of Patients with Severe Coronary Artery Calcification Undergoing Orbital Atherectomy. J Interv Cardiol. 2016 Aug;29(4):357-62. doi: 10.1111/joic.12310. Epub 2016 Jun 30. PMID 27358246
- [Background] Madhavan MV, Shahim B, Mena-Hurtado C, Garcia L, Crowley A, Parikh SA. Efficacy and safety of intravascular lithotripsy for the treatment of peripheral arterial disease: An individual patient-level pooled data analysis. Catheter Cardiovasc Interv. 2020 Apr 1;95(5):959-968. doi: 10.1002/ccd.28729. Epub 2020 Jan 20. PMID 31957955
- [Background] Madhavan MV, Tarigopula M, Mintz GS, Maehara A, Stone GW, Genereux P. Coronary artery calcification: pathogenesis and prognostic implications. J Am Coll Cardiol. 2014 May 6;63(17):1703-14. doi: 10.1016/j.jacc.2014.01.017. Epub 2014 Feb 12. PMID 24530667
- [Background] McClelland RL, Chung H, Detrano R, Post W, Kronmal RA. Distribution of coronary artery calcium by race, gender, and age: results from the Multi-Ethnic Study of Atherosclerosis (MESA). Circulation. 2006 Jan 3;113(1):30-7. doi: 10.1161/CIRCULATIONAHA.105.580696. Epub 2005 Dec 19. PMID 16365194
- [Background] Mintz GS. Intravascular imaging of coronary calcification and its clinical implications. JACC Cardiovasc Imaging. 2015 Apr;8(4):461-471. doi: 10.1016/j.jcmg.2015.02.003. PMID 25882575
- [Background] Mori H, Torii S, Kutyna M, Sakamoto A, Finn AV, Virmani R. Coronary Artery Calcification and its Progression: What Does it Really Mean? JACC Cardiovasc Imaging. 2018 Jan;11(1):127-142. doi: 10.1016/j.jcmg.2017.10.012. PMID 29301708
- [Background] Mori S, Yasuda S, Kataoka Y, Morii I, Kawamura A, Miyazaki S. Significant association of coronary artery calcification in stent delivery route with restenosis after sirolimus-eluting stent implantation. Circ J. 2009 Oct;73(10):1856-63. doi: 10.1253/circj.cj-09-0080. Epub 2009 Aug 27. PMID 19713655
- [Background] Nakahara T, Dweck MR, Narula N, Pisapia D, Narula J, Strauss HW. Coronary Artery Calcification: From Mechanism to Molecular Imaging. JACC Cardiovasc Imaging. 2017 May;10(5):582-593. doi: 10.1016/j.jcmg.2017.03.005. PMID 28473100
- [Background] Nakahara T, Narula J, Strauss HW. Calcification and Inflammation in Atherosclerosis: Which Is the Chicken, and Which Is the Egg? J Am Coll Cardiol. 2016 Jan 5;67(1):79-80. doi: 10.1016/j.jacc.2015.11.014. No abstract available. PMID 26764070
- [Background] Nakahara T, Strauss HW. From inflammation to calcification in atherosclerosis. Eur J Nucl Med Mol Imaging. 2017 May;44(5):858-860. doi: 10.1007/s00259-016-3608-x. No abstract available. PMID 28062896
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic' PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO. [2018 ESC/EACTS Guidelines on myocardial revascularization. The Task Force on myocardial revascularization of the European Society of Cardiology (ESC) and European Association for Cardio-Thoracic Surgery (EACTS)]. G Ital Cardiol (Rome). 2019 Jul-Aug;20(7-8 Suppl 1):1S-61S. doi: 10.1714/3203.31801. No abstract available. Italian. PMID 31379378
- [Background] Okura H, Hayase M, Shimodozono S, Kobayashi T, Sano K, Matsushita T, Kondo T, Kijima M, Nishikawa H, Kurogane H, Aizawa T, Hosokawa H, Suzuki T, Yamaguchi T, Bonneau HN, Yock PG, Fitzgerald PJ; REDUCE Investigators. Restenosis Reduction by Cutting Balloon Evaluation. Mechanisms of acute lumen gain following cutting balloon angioplasty in calcified and noncalcified lesions: an intravascular ultrasound study. Catheter Cardiovasc Interv. 2002 Dec;57(4):429-36. doi: 10.1002/ccd.10344. PMID 12455075
- [Background] Parikh K, Chandra P, Choksi N, Khanna P, Chambers J. Safety and feasibility of orbital atherectomy for the treatment of calcified coronary lesions: the ORBIT I trial. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1134-9. doi: 10.1002/ccd.24700. Epub 2013 Mar 5. PMID 23460596
- [Background] Raber L, Mintz GS, Koskinas KC, Johnson TW, Holm NR, Onuma Y, Radu MD, Joner M, Yu B, Jia H, Meneveau N, de la Torre Hernandez JM, Escaned J, Hill J, Prati F, Colombo A, Di Mario C, Regar E, Capodanno D, Wijns W, Byrne RA, Guagliumi G. Clinical use of intracoronary imaging. Part 1: guidance and optimization of coronary interventions. An expert consensus document of the European Association of Percutaneous Cardiovascular Interventions. EuroIntervention. 2018 Aug 20;14(6):656-677. doi: 10.4244/EIJY18M06_01. PMID 29939149
- [Background] Sangiorgi G, Rumberger JA, Severson A, Edwards WD, Gregoire J, Fitzpatrick LA, Schwartz RS. Arterial calcification and not lumen stenosis is highly correlated with atherosclerotic plaque burden in humans: a histologic study of 723 coronary artery segments using nondecalcifying methodology. J Am Coll Cardiol. 1998 Jan;31(1):126-33. doi: 10.1016/s0735-1097(97)00443-9. PMID 9426030
- [Background] Secco GG, Ghione M, Mattesini A, Dall'Ara G, Ghilencea L, Kilickesmez K, De Luca G, Fattori R, Parisi R, Marino PN, Lupi A, Foin N, Di Mario C. Very high-pressure dilatation for undilatable coronary lesions: indications and results with a new dedicated balloon. EuroIntervention. 2016 Jun 20;12(3):359-65. doi: 10.4244/EIJY15M06_04. PMID 26111405
- [Background] Sorini Dini C, Nardi G, Ristalli F, Mattesini A, Hamiti B, Di Mario C. Contemporary Approach to Heavily Calcified Coronary Lesions. Interv Cardiol. 2019 Nov 18;14(3):154-163. doi: 10.15420/icr.2019.19.R1. eCollection 2019 Nov. PMID 31867062
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Background] Tzafriri AR, Garcia-Polite F, Zani B, Stanley J, Muraj B, Knutson J, Kohler R, Markham P, Nikanorov A, Edelman ER. Calcified plaque modification alters local drug delivery in the treatment of peripheral atherosclerosis. J Control Release. 2017 Oct 28;264:203-210. doi: 10.1016/j.jconrel.2017.08.037. Epub 2017 Sep 1. PMID 28867375
- [Background] van Setten J, Isgum I, Smolonska J, Ripke S, de Jong PA, Oudkerk M, de Koning H, Lammers JW, Zanen P, Groen HJ, Boezen HM, Postma DS, Wijmenga C, Viergever MA, Mali WP, de Bakker PI. Genome-wide association study of coronary and aortic calcification implicates risk loci for coronary artery disease and myocardial infarction. Atherosclerosis. 2013 Jun;228(2):400-5. doi: 10.1016/j.atherosclerosis.2013.02.039. Epub 2013 Mar 13. PMID 23561647
- [Background] Wang X, Matsumura M, Mintz GS, Lee T, Zhang W, Cao Y, Fujino A, Lin Y, Usui E, Kanaji Y, Murai T, Yonetsu T, Kakuta T, Maehara A. In Vivo Calcium Detection by Comparing Optical Coherence Tomography, Intravascular Ultrasound, and Angiography. JACC Cardiovasc Imaging. 2017 Aug;10(8):869-879. doi: 10.1016/j.jcmg.2017.05.014. PMID 28797408
- [Background] Wiemer M, Butz T, Schmidt W, Schmitz KP, Horstkotte D, Langer C. Scanning electron microscopic analysis of different drug eluting stents after failed implantation: from nearly undamaged to major damaged polymers. Catheter Cardiovasc Interv. 2010 May 1;75(6):905-11. doi: 10.1002/ccd.22347. PMID 20088011
- [Background] Willemink MJ, Leiner T, Maurovich-Horvat P. Cardiac CT Imaging of Plaque Vulnerability: Hype or Hope? Curr Cardiol Rep. 2016 Apr;18(4):37. doi: 10.1007/s11886-016-0714-0. PMID 26922591
- [Background] Wong ND, Kouwabunpat D, Vo AN, Detrano RC, Eisenberg H, Goel M, Tobis JM. Coronary calcium and atherosclerosis by ultrafast computed tomography in asymptomatic men and women: relation to age and risk factors. Am Heart J. 1994 Feb;127(2):422-30. doi: 10.1016/0002-8703(94)90133-3. PMID 8296711
- [Background] Yamamoto H, Imazu M, Hattori Y, Tadehara F, Yamakido M, Nakanishi T, Ito K. Predicting angiographic narrowing > or = 50% in diameter in each of the three major arteries by amounts of calcium detected by electron beam computed tomographic scanning in patients with chest pain. Am J Cardiol. 1998 Mar 15;81(6):778-80. doi: 10.1016/s0002-9149(97)01011-4. PMID 9527093
- [Background] Yamamoto MH, Maehara A, Karimi Galougahi K, Mintz GS, Parviz Y, Kim SS, Koyama K, Amemiya K, Kim SY, Ishida M, Losquadro M, Kirtane AJ, Haag E, Sosa FA, Stone GW, Moses JW, Ochiai M, Shlofmitz RA, Ali ZA. Mechanisms of Orbital Versus Rotational Atherectomy Plaque Modification in Severely Calcified Lesions Assessed by Optical Coherence Tomography. JACC Cardiovasc Interv. 2017 Dec 26;10(24):2584-2586. doi: 10.1016/j.jcin.2017.09.031. No abstract available. PMID 29268891
- [Background] Yeoh J, Hill J. Intracoronary Lithotripsy for the Treatment of Calcified Plaque. Interv Cardiol Clin. 2019 Oct;8(4):411-424. doi: 10.1016/j.iccl.2019.06.004. PMID 31445725
- [Background] Zhang J, Gao X, Kan J, Ge Z, Han L, Lu S, Tian N, Lin S, Lu Q, Wu X, Li Q, Liu Z, Chen Y, Qian X, Wang J, Chai D, Chen C, Li X, Gogas BD, Pan T, Shan S, Ye F, Chen SL. Intravascular Ultrasound Versus Angiography-Guided Drug-Eluting Stent Implantation: The ULTIMATE Trial. J Am Coll Cardiol. 2018 Dec 18;72(24):3126-3137. doi: 10.1016/j.jacc.2018.09.013. Epub 2018 Sep 24. PMID 30261237